CLINICAL TRIAL: NCT01402479
Title: An Open-labeled Trial of Ramipril in Patients With Migraine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Manho Kim, MD, PhD, Department of Neurology, Seoul National University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0408-131-005
Record Dates: First submitted 2011-07-24; First posted 2011-07-26 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2011-07

CONDITIONS: Migraine With Hypertension
Keywords: migraine,; ramipril,; hypertension
MeSH Terms: conditions — Migraine Disorders; Hypertension | interventions — Ramipril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ramipril (Active Comparator): open label single arm trial
  Interventions: Drug: Ramipril

INTERVENTIONS:
Drug: Ramipril — ramipril 2.5mg twice a day

SUMMARY:
Physiology of migraine involving renin-angiotensin systems (RAS) has been implicated. Ramipril is a broadly-used angiotensin-converting enzyme inhibitor. The investigators attempt to test the efficacy of ramipril on the prophylaxis of migraine attacks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic migraine are included in this study. Migraineurs should be aged 20 to 70 years old with the ability to read and understand the self-report scales, including the headache diary, used in this study.

Exclusion Criteria:

1. Medication overuse headache are excluded in this study.
2. Treatment with other ACEI or medication that may affect ARS
3. Treatment with migraine prophylactic medications or anti-hypertensive agents including β adrenergic receptor or calcium channel blockers
4. Past history of hepatic or renal dysfunction; an abnormal electrocardiography; a psychiatric disorder; a history of substance abuse; pregnancy or lactation; use of anti-psychotics, antidepressants, or anti-anxiety drugs.

Ages: 20 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2004-10; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
headache frequency | 12 week
  headache days

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea